CLINICAL TRIAL: NCT04610008
Title: Optic Nerve Head Shape as a Predictor of the Formation of Acquired Pits of the Optic Nerve (APONs)
Status: Completed | Type: Observational
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Other Study IDs: 7943
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2020-10

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- APON: Retrospective review of routine clinical images from patients with an acquired pit of the optic nerve (APON), and a documented diagnosis of primary open angle glaucoma or normal tension glaucoma
  Interventions: Other: No intervention. Purely observation
- No APON control: Retrospective review of routine clinical images from patients with NO acquired pit of the optic nerve (APON), and a documented diagnosis of primary open angle glaucoma or normal tension glaucoma
  Interventions: Other: No intervention. Purely observation

INTERVENTIONS:
Other: No intervention. Purely observation — Retrospective image analysis of the shape of the optic nerve head in both groups

SUMMARY:
Acquired pits of the optic nerve (APONs) are an area of focal loss of neural tissue associated with a discrete area of depression/excavation within the optic cup at the level of the lamina cribrosa. It is commonly associated with glaucoma and can be seen on the optic disc when examining the back of a patient's eye. It causes a characteristic visual field defect in the central 5-10 degrees of vision which has a significant impact of a patient's daily activities. There is no treatment to restore vision once it has formed.

Previous studies suggest mechanical stress across this part of the eye may have role in the formation of APONs. The investigators therefore hypothesise that if a patient has a more elliptical shaped optic disc, which would have more irregular mechanical stress across it, it may have a higher risk of an APON forming.

Patients with glaucoma attending the ophthalmology department at University Hospital of Wales have regular photographs taken of the optic nerve/optic disc as part of their routine clinical care in order to monitor the condition. The research team, who are all practicing ophthalmologists in the department, will review anonymised photographs to find optic discs with APONs, and another group with glaucoma but no APONs to use as a control. The research team will then measure the dimensions of the optic disc to determine if APONs are more common in optic discs with a more elliptical shape. The patients' clinical notes will then need to be accessed to collect data on the age, sex and diagnosis. This data will be anonymised using ID numbers once collected.

The final outcomes of the study will the average measured dimensions of the optic disc in each group, and the position that the APON occurs.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of primary open angle glaucoma (POAG) or normal tension glaucoma (NTG)
* Under the care of the ophthalmology department at University Hospital of Wales
* Available optic disc photograph
* Presence of an APON for disease group, no APON for control group

Exclusion Criteria:

* No documented diagnosis of POAG/NTG
* Other form of glaucoma - e.g. traumatic glaucoma/juvenile glaucoma
* Poor photograph quality
* Optic disc tilted so that the margin is obscured and cannot be demarcated
* Coexisting disc pathology, e.g. congenital optic disc pit

Ages: 50 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients under the care of University Hospital of Wales Ophthalmology Department with optic nerve head photographs taken as part of routine clinical care for monitoring of glaucoma.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Optic disc radius ratio | 6 months
  Comparison of the ratio of the maximum/minimum optic disc radius for optic discs with APONs and optic discs with glaucoma but no APON.

SECONDARY OUTCOMES:
The percentile rank of the disc radius at the position of the APON | 6 months
  The percentile rank of the disc radius at the position of the APON

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Wales, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No